CLINICAL TRIAL: NCT01802346
Title: A Randomized, Phase II Clinical Trial of a Controlled Diet Prior to Selected Chemotherapy Treatment in Breast and Prostate Cancer to Evaluate the Impact on Toxicity and Efficacy
Brief Title: Controlled Low Calorie Diet in Reducing Side Effects and Increasing Response to Chemotherapy in Patients With Breast or Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-10-3; NCI-2013-00414 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Diet Therapy; Nutritional Support; Nutrition Assessment; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (low-calorie diet) (Experimental): Patients eat a special low-calorie diet during 3 days prior to chemotherapy, during the 12 weeks of chemotherapy, and 2 days after chemotherapy. Patients are provided with all meals and all food to be consumed and maintain a diary of the food consumed and appropriate amounts.
  Interventions: Dietary Supplement: dietary intervention; Other: laboratory biomarker analysis
- Arm II (normal diet) (Active Comparator): Patients eat a normal diet and receive dietary advice which may include consultation with a nutritionist. Patients maintain a diary of the food consumed and appropriate amounts.
  Interventions: Procedure: nutritional support; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: dietary intervention — Consume a low-calorie diet
  Other Names: Dietary Modification; intervention, dietary
  Arms: Arm I (low-calorie diet)
Procedure: nutritional support — Receive dietary advice
  Other Names: nutritional assessment; nutritional care; support, nutritional
  Arms: Arm II (normal diet)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well a controlled low calorie diet works in reducing side effects and increasing response to chemotherapy in patients with breast or prostate cancer. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Eating a special diet with low calories may reduce the side effects of chemotherapy and improve the response to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary estimates of the impact of a restricted diet on toxicity and efficacy of chemotherapy for breast and prostate cancer.

II. To evaluate the compliance with a controlled diet intervention.

III. To investigate changes in plasma insulin, glucose, insulin-like growth factor 1 (IGF1) and IGF binding protein (IGFBP) levels in subjects who consume a restricted diet compared to controls.

OUTLINE:

Patients are randomized to 1 or 2 treatment arms.

ARM I: Patients eat a special low-calorie diet during 3 days prior to chemotherapy, during the 12 weeks of chemotherapy, and 24 hours after chemotherapy. Patients are provided with all meals and all food to be consumed and maintain a diary of the food consumed and appropriate amounts. Patients meet with the study dietician within 3 weeks of enrollment and prior to, or on the day of, their first course of chemotherapy on study and at the start of each subsequent course.

ARM II: Patients eat a normal diet and receive dietary advice which may include consultation with a nutritionist. Patients maintain a diary of the food consumed and appropriate amounts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer for which chemotherapy with AC (doxorubicin plus cyclophosphamide) is being utilized in the neoadjuvant or adjuvant setting OR metastatic prostate adenocarcinoma for which Docetaxel will be administered
* Body mass index (BMI) >= 18.5
* Subjects do not need to have measurable or evaluable disease; chemotherapy may be administered in the neoadjuvant, adjuvant, or metastatic setting
* Prior therapy:

  * Breast cancer subjects may not have received prior chemotherapy, with the exception of curative-intent chemotherapy for a separate malignancy more than 3 years ago
  * Prostate cancer subjects may have received prior treatment with metronomic cyclophosphamide as this is considered anti-angiogenic/immunomodulatory and not cytotoxic
  * Prostate cancer subjects may be receiving a 2nd course of docetaxel provided that ** The first course resulted in a PSA response (> 30% reduction in prostate specific antigen [PSA] and/or improvement in radiographic findings or pain) and the last dose was >= 9 months ago
* Prior Radiotherapy is allowed, provided at least 2 weeks have elapsed from completion of radiotherapy to initiation of protocol treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2x upper limit of normal (ULN)
* Absolute neutrophil count (ANC) > 1500
* Platelets (plts) > 90,000
* Premenopausal women must have a negative pregnancy test and must agree to use barrier contraception throughout the study period

Exclusion Criteria:

* Diabetes Mellitus
* Peripheral Neuropathy >= grade 1
* Prior therapy with inhibitors of IGF-1
* Concurrent use of somatostatin
* Significant food allergies which would make the subject unable to consume the food provided (ex: shellfish, soy or egg allergy)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2027-06-29 (Estimated)

PRIMARY OUTCOMES:
Rate of chemotherapy-related toxicity | Up to 12 weeks
  Occurrence of Grade 2+ non-hematologic symptomatic toxicity (fatigue, nausea and vomiting, anorexia, neuropathy, mucositis, cystitis, stomatitis), evaluated according to Common Terminology Criteria for Adverse Events version 4.0. The two arms will be compared, in terms of the proportion of patients with the occurrence of one of these toxicities.

SECONDARY OUTCOMES:
Tumor response | Up to 12 weeks
  Measured using a summary statistic which includes Response Evaluation Criteria In Solid Tumors (RECIST) response, PSA response for men without measurable disease, pathologic complete response and clinical response for breast cancer patients. This rate will be compared between patients on the restricted diet and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Spicer, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Mayo Clinic Rochester, Rochester, Minnesota